CLINICAL TRIAL: NCT02268383
Title: An Open-Label Extension Study to Evaluate the Long-Term Effects of ACE-536 for the Treatment of Anemia in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndromes (MDS) Previously Enrolled in Study A536-03
Brief Title: Extension Study to Evaluate Long-Term Effects of Luspatercept in Patients With Myelodysplastic Syndromes (MDS) (A536-05/MK-6143-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A536-05; MK-6143-003 (Other: Merck); A536-05 (Other: Acceleron); 2014-001280-13 (EudraCT Number)
Record Dates: First submitted 2014-10-06; First posted 2014-10-20 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Luspatercept Extension population (Experimental): Luspatercept 1.0 mg/kg once every 3 weeks by subcutaneous injection.
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Luspatercept 1.0 mg/kg once every 3 weeks by subcutaneous injection.
  Other Names: MK-6143; ACE-536

SUMMARY:
This study is an open-label extension study for participants previously enrolled in study MK-6143-001 (formerly called A536-03, ClinicalTrials.gov Identifier NCT01749514), to evaluate the long-term safety and tolerability of luspatercept (MK-6143) in participants with low or intermediate-1 risk MDS.

DETAILED DESCRIPTION:
This study is an open-label extension study to evaluate the safety, tolerability, and pharmacodynamic effects of up to 24 months of luspatercept treatment in participants with low or intermediate-1 risk myelodysplastic syndromes previously treated with luspatercept for up to 3 months in MK-6143-001 study (NCT01749514). The starting dose level in this study will be 1.0 mg/kg by subcutaneous (SC) injection every 3 weeks. Dose titration/modification rules will be followed for individual participants and will be based upon safety and efficacy data collected during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the treatment period in the base study MK-6143-001 (ClinicalTrials.gov Identifier: NCT01749514)
* Adequate birth control measures
* Patient is able to adhere to the study visit schedule, understand and comply with all protocol requirements
* Patient understands and is able to provide written informed consent
* In addition, patients with treatment interruption (defined as patients who complete their end-of-study visit in MK-6143-001 and cannot directly roll over to MK-6143-003) must also meet the following criteria:

  * Documented diagnosis of idiopathic/de novo MDS or non-proliferative chronic myelomonocytic leukemia (CMML) according to the World Health Organization (WHO) criteria 16 (white blood count (WBC) < 13,000/μL) that meets International Prognostic Scoring System (IPSS) classification of low or intermediate-1 risk disease as determined by microscopic and standard cytogenetic analyses of the bone marrow and peripheral complete blood count (CBC) obtained during screening;
* Anemia defined as:

  * Mean hemoglobin concentration < 10.0 g/dL of 2 measurements (one performed within one day prior to Cycle 1 Day 1 and the other performed 7-28 days prior to Cycle 1 Day 1), for non-transfusion dependent (NTD) patients (defined as having received ˂ 4 units of red blood cells (RBCs) within 8 weeks prior to Cycle 1 Day 1), OR
  * Transfusion Dependent (TD), defined as having received ≥ 4 units of RBCs within 8 weeks prior to Cycle 1 Day 1
* Platelet count ≥ 30 x 109/L
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (if related to anemia)
* Adequate renal (creatinine ≤ 2.0 x upper limit of normal [ULN]) and hepatic (total bilirubin < 2 x ULN and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN) function

Exclusion Criteria:

* Discontinuation/withdrawal from the base study A536-03 (due to patient request, patient unwillingness or inability to comply with the protocol, pregnancy, use of prohibited medication [e.g. azacitidine], medical reason or adverse event (AE), hypersensitivity reaction to the study drug, at the discretion of the sponsor, or loss to follow-up) prior to completion of the treatment period
* Prior treatment with azacitidine or decitabine
* Treatment within 28 days prior to Cycle 1 Day 1 with:

  * An erythropoiesis-stimulating agent (ESA),
  * Granulocyte colony-stimulating factor (G-CSF) and granulocyte-macrophage colony stimulating factor (GM-CSF),
  * Lenalidomide
* Iron chelation therapy if initiated within 56 days prior to Cycle 1 Day 1
* Treatment with another investigational drug (including sotatercept [ACE-011]) or device, or approved therapy for investigational use ≤ 28 days prior to Cycle 1 Day 1, or if the half-life of the previous investigational product is known, within 5 times the half-life prior to Cycle 1 Day 1, whichever is longer
* Major surgery within 28 days prior to Cycle 1 Day 1. Patients must have completely recovered from any previous surgery prior to Cycle 1 Day 1
* Known positive for human immunodeficiency virus (HIV), active infectious hepatitis B (HBV) or active infectious hepatitis C (HCV)
* Uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 150 mm Hg or diastolic blood pressure (DBP) ≥ 100 mm Hg
* Pregnant or lactating females
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational drug
* Any other condition not specifically noted above which, in the judgment of the investigator, would preclude the patient from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Acceleron Investigative Site, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Platzbecker U, Gotze KS, Kiewe P, Germing U, Mayer K, Radsak M, Wolff T, Chromik J, Sockel K, Oelschlagel U, Haase D, Illmer T, Al-Ali HK, Silling G, Reynolds JG, Zhang X, Attie KM, Shetty JK, Giagounidis A. Long-Term Efficacy and Safety of Luspatercept for Anemia Treatment in Patients With Lower-Risk Myelodysplastic Syndromes: The Phase II PACE-MDS Study. J Clin Oncol. 2022 Nov 20;40(33):3800-3807. doi: 10.1200/JCO.21.02476. Epub 2022 Aug 23. PMID 35998303
- [Derived] Platzbecker U, Germing U, Gotze KS, Kiewe P, Mayer K, Chromik J, Radsak M, Wolff T, Zhang X, Laadem A, Sherman ML, Attie KM, Giagounidis A. Luspatercept for the treatment of anaemia in patients with lower-risk myelodysplastic syndromes (PACE-MDS): a multicentre, open-label phase 2 dose-finding study with long-term extension study. Lancet Oncol. 2017 Oct;18(10):1338-1347. doi: 10.1016/S1470-2045(17)30615-0. Epub 2017 Sep 1. PMID 28870615

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This extension study enrolled participants from base study MK-6143-001 (NCT01749514). Participants were referred as 'Direct Roll Over' participants (n=67; enrolled within ~28 days after last dose of luspatercept and did not complete post treatment follow up (PTFU) or end of study (EOS) visit of base study) or 'Treatment Interrupted' participants (n=8; completed EOS visit for base study). Per protocol, a total of 75 participants were pooled together in the extension study.
Groups:
- Luspatercept Extension Population: Participants received luspatercept dose of either 0.5, 0.75, 1.0, 1.33, or 1.75 mg/kg determined via Fibonacci scheme on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years) as a subcutaneous (SC) injection. Direct Roll Over participants received the highest tolerated dose of luspatercept that was assigned in the base study. Treatment Interrupted participants received an initial dose of luspatercept 1mg/kg on Day 1 of Cycle 1 (cycle length = 21 days) and the subsequent doses were titrated up to 1.75mg/kg Q3W via Fibonacci scheme, on Day 1 of each cycle for up to 87 cycles (for up to approximately 5 years).
Period: Overall Study
Arm/Group | Luspatercept Extension Population
Started | 75
Completed | 14
Not Completed | 61
Not completed — Death | 12
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 9
Not completed — Presence of ≥1% blasts in peripheral blood | 1
Not completed — Protocol deviation | 3
Not completed — Sponsor decision | 22
Not completed — Not reported | 12

BASELINE CHARACTERISTICS:
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0
Transfusion Status [Count of Participants; unit: Participants] — Low Transfusion Burden (LTB) participants are defined as those who received < 4 units of red blood cells (RBCs) within 8 weeks prior to baseline (Cycle 1 Day 1). High Transfusion Burden (HTB) participants are defined as those who required ≥4 units of RBC transfusions within 8 weeks prior to baseline.
  Participants
    HTB | 25
    LTB | 50
Hemoglobin level [Mean (Standard Deviation); unit: grams/dl] — Hemoglobin level of participants in peripheral blood at baseline was reported. Population: All enrolled participants with baseline hemoglobin level data available. Data were not collected from 2 participants at baseline.
  grams/dl
    number analyzed (Participants) | 73
    (all) | 8.74 (1.01)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who experienced an AE was reported.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who received at least one dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 75
Participants | 75

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who discontinued luspatercept due to an AE was reported.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who received at least one dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 75
Participants | 23

3. Secondary Outcome: Percentage of Participants With Modified Erythroid Response (mHI-E) Per International Working Group (IWG) 2006 Response Criteria
Description: The mHI-E was defined as a mean hemoglobin (Hgb) increase ≥1.5 g/dL over an 8-week period as compared to baseline, not influenced by red blood cell (RBC) transfusion in low transfusion burden (LTB) participants and a decrease of ≥4 units or ≥50% of units of RBCs transfused over a period of 8 weeks, relative to the number of units of RBCs transfused in the 8 weeks immediately prior to baseline in high transfusion burden (HTB) participants. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. HTB participants were those who required a transfusion of ≥4 units of RBCs in the 8 weeks prior to baseline. Rolling 8 weeks was defined as any consecutive 8 weeks during the study.
Time Frame: Any consecutive 8 weeks during the study (up to approximately 5 years)
Population: All enrolled participants who received at least one dose of luspatercept and were mHI-E evaluable.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 75
Percentage of participants | 81.3 [70.7 to 89.4]

4. Secondary Outcome: Rate of Erythroid Response (HI-E) Per IWG 2006 Response Criteria
Description: Per IWG 2006 response criteria, the rate of HI-E was defined as the percentage of participants with an HI-E response by an Hgb increase of ≥1.5 g/dL for participants not transfused or as defined by having received less than 4 units of RBCs within 8 weeks of baseline or reduction by ≥4 units of RBCs transfused (for a Hgb≤9.0 g/dL) during any 8-week period on study, compared with the 8-week period prior to study day 1.
Time Frame: Any consecutive 8 weeks during the study (up to approximately 5 years)
Population: All enrolled participants who received at least one dose of luspatercept and were HI-E evaluable.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 75
Percentage of participants | 80.0 [69.2 to 88.4]

5. Secondary Outcome: Rate of Neutrophil Response (HI-N) Per IWG 2006 Response Criteria
Description: Per IWG 2006 response criteria, HI-N response was defined for participants with baseline absolute neutrophil count (ANC) <1.0×10^9/L as the percentage increase ≥100% and an absolute mean increase >0.5 ×10^9/L during any rolling 8-week window on treatment compared with baseline. The rolling 8-week was defined as any consecutive 8 weeks during the study. Percentage of participants with HI-N response were reported.
Time Frame: Any consecutive 8 Weeks during the study (up to approximately 5 years)
Population: All enrolled participants who received at least one dose of luspatercept and had baseline neutrophil count <1.0×10^9/L.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 14
Percentage of participants | 64.3 [35.1 to 87.2]

6. Secondary Outcome: Rate of Platelet Response (HI-P) Per IWG 2006 Response Criteria
Description: Per IWG 2006 response criteria, HI-P response was defined for participants with baseline platelet count <100×10^9/L as the following: 1) For participants with baseline ≥20×10^9/L, an absolute increase of ≥30×10^9/L during any rolling 8-week window on treatment and 2) For participants with baseline <20×10^9/L, mean value of >20×10^9/L and percentage increase ≥100% during any rolling 8-week window on treatment. The rolling 8-week was defined as any consecutive 8 weeks during the study. Percentage of participants with HI-P response were reported.
Time Frame: Any consecutive 8 Weeks during the study (up to approximately 5 years)
Population: All enrolled participants who received at least one dose of luspatercept and had baseline platelet <100x10^9/L.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 11
Percentage of participants | 36.4 [10.9 to 69.2]

7. Secondary Outcome: Duration of HI-E in LTB Participants Per IWG 2006 Response Criteria
Description: For LTB participants, HI-E was defined as all Hgb increase ≥1.5 g/dL during any rolling 8 weeks window. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. Per IWG 2006 response criteria, duration of HI-E was defined as the time from the first day of the first rolling 8 weeks interval of showing response to the last day of the last consecutive rolling 8 weeks interval of showing response. Rolling 8 weeks was defined as any consecutive 8 weeks during the study. When there were multiple disjointed intervals with response, the longest interval was used.
Time Frame: up to approximately 5 years
Population: All enrolled LTB participants who received at least one dose of luspatercept and had a HI-E.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 50
Days | 299 (378.3)

8. Secondary Outcome: Duration of HI-E in HTB Participants Per IWG 2006 Response Criteria
Description: For HTB participants, HI-E was defined as RBC transfusion reduction ≥4 units during any rolling 8 weeks. HTB participants were those who required a transfusion of ≥4 units of RBCs in the 8 weeks prior to baseline. Per IWG 2006 response criteria, duration of HI-E was defined as the time from the first day of the first rolling 8 weeks interval of showing response to the last day of the last consecutive rolling 8 weeks interval of showing response. Rolling 8 weeks was defined as any consecutive 8 weeks during the study. When there were multiple disjointed intervals with response, the longest interval was used.
Time Frame: up to approximately 5 years
Population: All enrolled HTB participants who received at lease one dose of luspatercept and had a HI-E.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 25
Days | 328 (286.8)

9. Secondary Outcome: Time to HI-E in LTB Participants Per IWG 2006 Response Criteria
Description: For LTB participants, HI-E was defined as all Hgb increase ≥1.5 g/dL during any rolling 8 weeks window. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. Per IWG 2006 response criteria, time to HI-E was defined as the first date of the rolling 8 weeks interval of showing response minus first dose date plus 1. Rolling 8 weeks was defined as any consecutive 8 weeks during the study. When there were multiple disjointed intervals with response, the longest interval was used.
Time Frame: up to approximately 5 years
Population: All enrolled LTB participants who received at least one dose of luspatercept and had a HI-E.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 50
Days | 83 (86.2)

10. Secondary Outcome: Time to HI-E in HTB Participants Per IWG 2006 Response Criteria
Description: For HTB participants, HI-E was defined as RBC transfusion reduction ≥4 units during any rolling 8 weeks. HTB participants were those who required a transfusion of ≥4 units of RBCs in the 8 weeks prior to baseline. Per IWG 2006 response criteria, time to HI-E was defined as the first date of the rolling 8 weeks interval of showing response minus first dose date plus 1. Rolling 8 weeks was defined as any consecutive 8 weeks during the study.
Time Frame: Any consecutive 8 weeks during the study (up to approximately 5 years)
Population: All enrolled HTB participants who received at lease one dose of luspatercept and had a HI-E.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 25
Days | 13 (22.6)

11. Secondary Outcome: Rate of RBC Transfusion Independence (RBC-TI)
Description: Per protocol, RBC-TI response was defined as not requiring RBC transfusion for 8 or more weeks while on treatment among participants with ≥2 units of RBC transfusions at baseline. The rate of RBC-TI was defined as the percentage of participants with ≥2 units of RBC transfusions at baseline with RBC-TI.
Time Frame: Any consecutive 8 Weeks during the study (up to approximately 5 years)
Population: All enrolled participants who received at least one dose of luspatercept and had ≥2 units of RBC transfusions at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 42
Percentage of participants | 64.3 [48.0 to 78.4]

12. Secondary Outcome: Mean Change From Baseline to Week 8 in RBC Transfusion Burden (TB) in HTB Participants
Description: RBC TB was defined as ≥4 units or 50% reduction during rolling 8 weeks among HTB participants. The rolling 8-week was defined as any consecutive 8 weeks during the study. HTB participants are those who required a transfusion of ≥4 units of RBCs in the 8 weeks prior to baseline. Mean change from baseline to Week 8 in reduction in RBC TD in HTB participants was reported.
Time Frame: Baseline and up to 5 years
Population: All enrolled HTB participants who received at least one dose of luspatercept.
Measure: Mean (Standard Deviation); unit: Units of blood
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 25
Units of blood | -4.4 (2.6)

13. Secondary Outcome: Mean Change From Baseline to Week 8 in Hemoglobin Levels ≥1.5 Grams/dL in LTB Participants
Description: Baseline hemoglobin levels were the documented pre-transfusion hemoglobin values during the 12 weeks prior to treatment. LTB participants were those who received <4 units of RBCs within 8 weeks prior to baseline. Mean change from baseline to Week 8 in hemoglobin levels ≥1.5 grams/dL in LTB participants were reported.
Time Frame: Baseline and Week 8
Population: All enrolled LTB participants who received at least one dose of luspatercept.
Measure: Mean (Standard Deviation); unit: grams/dl
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 50
grams/dl | 2.4 (1.0)

14. Secondary Outcome: Serum Concentration of Luspatercept
Description: Blood samples were collected at pre-determined time points to determine the serum concentration of luspatercept. Serum concentrations that were below the limit of quantitation (LOQ) of the assay prior to the first dose were assigned a numerical value of zero. Post-treatment serum concentrations that were below the LOQ of the assay were treated as missing. Serum concentrations assigned a value of missing were omitted from the analysis. The LOQ of the assay was 50 ng/mL.
Time Frame: Day 1: Cycles 1, 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, and 81 (each cycle length = 21 days); End of treatment (EOT) Day 1853
Population: All participants who received at least one dose of luspatercept and had data available for serum concentration analysis available at each time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 55
µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 14
  Cycle 1 Day 1 | 0.509 (0.738)
  Cycle 5 Day 1: number analyzed (Participants) | 33
  Cycle 5 Day 1 | 6.373 (3.527)
  Cycle 9 Day 1 | 6.589 (4.32)
  Cycle 13 Day 1: number analyzed (Participants) | 33
  Cycle 13 Day 1 | 7.154 (4.423)
  Cycle 17 Day 1: number analyzed (Participants) | 38
  Cycle 17 Day 1 | 8.136 (4.476)
  Cycle 21 Day 1: number analyzed (Participants) | 33
  Cycle 21 Day 1 | 8.227 (3.811)
  Cycle 25 Day 1: number analyzed (Participants) | 31
  Cycle 25 Day 1 | 7.986 (4.061)
  Cycle 29 Day 1: number analyzed (Participants) | 28
  Cycle 29 Day 1 | 8.379 (2.884)
  Cycle 33 Day 1: number analyzed (Participants) | 25
  Cycle 33 Day 1 | 8.024 (3.035)
  Cycle 37 Day 1: number analyzed (Participants) | 22
  Cycle 37 Day 1 | 8.017 (3.724)
  Cycle 41 Day 1: number analyzed (Participants) | 17
  Cycle 41 Day 1 | 7.559 (3.582)
  Cycle 45 Day 1: number analyzed (Participants) | 13
  Cycle 45 Day 1 | 8.614 (4.015)
  Cycle 49 Day 1: number analyzed (Participants) | 12
  Cycle 49 Day 1 | 9.447 (2.967)
  Cycle 53 Day 1: number analyzed (Participants) | 10
  Cycle 53 Day 1 | 7.936 (2.982)
  Cycle 57 Day 1: number analyzed (Participants) | 8
  Cycle 57 Day 1 | 8.891 (3.053)
  Cycle 61 Day 1: number analyzed (Participants) | 6
  Cycle 61 Day 1 | 8.288 (3.753)
  Cycle 65 Day 1: number analyzed (Participants) | 4
  Cycle 65 Day 1 | 8.698 (4.729)
  Cycle 69 Day 1: number analyzed (Participants) | 4
  Cycle 69 Day 1 | 7.603 (3.144)
  Cycle 73 Day 1: number analyzed (Participants) | 4
  Cycle 73 Day 1 | 8.559 (3.68)
  Cycle 77 Day 1: number analyzed (Participants) | 4
  Cycle 77 Day 1 | 7.539 (2.555)
  Cycle 81 Day 1: number analyzed (Participants) | 1
  Cycle 81 Day 1 | 9.837 (NA) — NA = SD could not be calculated due to low number of participants with serum concentration of luspatercept.
  EOT (Day 1853): number analyzed (Participants) | 49
  EOT (Day 1853) | 6.732 (4.356)

15. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Serum Iron
Description: Blood samples were collected at pre-specified time intervals to determine serum iron concentration. The percentage change from baseline to Day 1853 in concentration of serum iron was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for serum iron.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 55
Percent change | 20.38 (70.489)

16. Secondary Outcome: Percent Change From Baseline to Day 1853 in Total Iron Binding Capacity (TIBC)
Description: Blood samples were collected at pre-specified time intervals to determine TIBC. The percentage change from baseline to Day 1853 in TIBC was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for TIBC.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 55
Percent change | -11.37 (11.979)

17. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Transferrin
Description: Blood samples were collected at pre-specified time intervals to determine serum transferrin concentration. The percentage change from baseline to Day 1853 in concentration of transferrin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for transferrin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 55
Percent change | -11.34 (11.587)

18. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Soluble Transferrin Receptor
Description: Blood samples were collected at pre-specified time intervals to determine soluble transferrin receptor concentration. The percentage change from baseline to Day 1853 in concentration of soluble transferrin receptor was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for soluble transferrin receptor.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 55
Percent change | 11.52 (48.541)

19. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Serum Ferritin
Description: Blood samples were collected at pre-specified time intervals to determine serum ferritin concentration. The percentage change from baseline to Day 1853 in concentration of serum ferritin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for serum ferritin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 55
Percent change | 71.61 (152.948)

20. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Non-Transferrin Bound Iron (NTBI)
Description: Blood samples were to be collected at pre-specified time intervals to determine concentration of NTBI. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: No data were collected for the percent change from baseline to day 1853 in concentration of NTBI.
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 0

21. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Serum Hepcidin
Description: Blood samples were to be collected at pre-specified time intervals to determine concentration of serum hepcidin. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: No data were collected for the percent change from baseline to day 1853 in concentration of serum hepcidin.
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 0

22. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Serum Erythropoietin
Description: Blood samples were collected at pre-specified time intervals to determine serum erythropoietin concentration. The percentage change from baseline to Day 1853 in concentration of serum erythropoietin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for erythropoietin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 53
Percent change | 2252.15 (14490.300)

23. Secondary Outcome: Percent Change From Baseline to Day 1853 in Reticulocyte Count
Description: Blood samples were collected at pre-specified time intervals to determine reticulocyte count. The percentage change from baseline to Day 1853 in reticulocyte count was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for reticulocyte.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 47
Percent change | 78.70 (137.168)

24. Secondary Outcome: Percent Change From Baseline to Day 1853 in Nucleated RBC (nRBC) Count
Description: Blood samples were to be collected at pre-specified time intervals to determine nRBC. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: No data were collected for the percent change from baseline to day 1853 in nRBC count.
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 0

25. Secondary Outcome: Percent Change From Baseline to Day 1853 in Direct Bilirubin Level
Description: Blood samples were collected at pre-specified time intervals to determine serum direct bilirubin concentration. The percentage change from baseline to Day 1853 in concentration of direct bilirubin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for direct bilirubin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 47
Percent change | 110.53 (572.494)

26. Secondary Outcome: Percent Change From Baseline to Day 1853 in Total Bilirubin Level
Description: Blood samples were collected at pre-specified time intervals to determine total bilirubin concentration. The percentage change from baseline to Day 1853 in concentration of total bilirubin was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for total bilirubin.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 57
Percent change | 72.17 (236.953)

27. Secondary Outcome: Percent Change From Baseline to Day 1853 in Lactate Dehydrogenase Level
Description: Blood samples were collected at pre-specified time intervals to determine serum lactate dehydrogenase level. The percentage change from baseline to Day 1853 in concentration of lactate dehydrogenase level was reported.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: All enrolled participants who received at least one dose of luspatercept and had data available for lactate dehydrogenase.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 55
Percent change | 22.98 (43.017)

28. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Serum Bone-Specific Alkaline Phosphatase (BSAP)
Description: Blood samples were to be collected at pre-specified time intervals to determine BSAP. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: No data were collected for the percent change from baseline to day 1853 in concentration of BSAP.
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 0

29. Secondary Outcome: Percent Change From Baseline to Day 1853 in Concentration of Serum Cross-Linked C-Telopeptide of Type I Collagen (CTX)
Description: Blood samples were to be collected at pre-specified time intervals to determine CTX. Baseline was prespecified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of luspatercept) and Day 1853
Population: No data were collected for the percent change from baseline to day 1853 in concentration of CTX.
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to approximately 5 years
Description: All-cause mortality was reported on all enrolled participants. Serious and non-serious adverse events were reported on all participants who received at least one dose of luspatercept. Data are presented by the dose of luspatercept that was administered at the time when the AE or death occurred.
Groups:
- Luspatercept 0.5 mg/kg: Participants received luspatercept dose of 0.5 mg/kg on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
- Luspatercept 0.75 mg/kg: Participants received luspatercept dose of 0.75 mg/kg on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
- Luspatercept 1 mg/kg: Participants received luspatercept dose of 1 mg/kg on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
- Luspatercept 1.33 mg/kg: Participants received luspatercept dose of 1.33 mg/kg on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
- Luspatercept 1.75 mg/kg: Participants received luspatercept dose of 1.75 mg/kg on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
Arm/Group | Luspatercept 0.5 mg/kg | Luspatercept 0.75 mg/kg | Luspatercept 1 mg/kg | Luspatercept 1.33 mg/kg | Luspatercept 1.75 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 4/73 | 3/61 | 6/49
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/2 | 19/73 | 16/61 | 34/49
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 44/73 | 29/61 | 38/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.5 mg/kg (N=1) | Luspatercept 0.75 mg/kg (N=2) | Luspatercept 1 mg/kg (N=73) | Luspatercept 1.33 mg/kg (N=61) | Luspatercept 1.75 mg/kg (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Autoinflammatory disease (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.5 mg/kg (N=1) | Luspatercept 0.75 mg/kg (N=2) | Luspatercept 1 mg/kg (N=73) | Luspatercept 1.33 mg/kg (N=61) | Luspatercept 1.75 mg/kg (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 5 (5)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (12)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (2) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (8) | 3 (6) | 7 (9)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 8 (9) | 2 (3) | 6 (8)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 7 (10) | 3 (3) | 8 (14)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 2 (4) | 4 (7)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 3 (11) | 4 (7) | 3 (5)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 10 (18)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 13 (18) | 5 (7) | 10 (16)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 6 (8)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 3 (6) | 3 (6) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (5) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (5) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 5 (13) | 1 (1) | 5 (6)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (6) | 5 (6) | 7 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 5 (10) | 2 (2) | 3 (8)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 3 (3)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 18 (31) | 5 (6) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abscess limb (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or disclosure of study results will be permitted except as specified in a separate, written, agreement between the sponsor and the investigator(s).

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT02268383/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT02268383/SAP_001.pdf